CLINICAL TRIAL: NCT02092714
Title: A Pilot Study Utilizing Molecular Analysis Via Cancer CodeTM to Identify Therapeutic Targets for Patients With Advanced Neuroendocrine Tumors
Brief Title: Molecular Analysis in Tissue Samples From Patients With Advanced or Metastatic Neuroendocrine Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CGI-061; NCI-2013-01950 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-040 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and tumor tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ancillary-correlative (molecular analysis): Previously collected tissue samples are analyzed via mutational sequencing and immunohistochemistry.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot research trial studies molecular analysis in tissue samples from patients with advanced or metastatic neuroendocrine tumors. Studying samples of tissue from patients with neuroendocrine tumors in the lab may help doctors identify mutations to classify disease and plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform gene panel sequencing of patients with neuroendocrine tumors under care at Fox Chase Cancer Center for the purpose of identifying therapeutic targets and prognostic markers.

II. To assess the feasibility of performing a clinical trial of molecularly matched therapy in patients with differing subtypes of neuroendocrine tumors (neuroendocrine tumors of the pancreas [PNETs], non-pancreatic neuroendocrine tumors [NETs], and poorly differentiated NETs), based upon the proportion of patients with actionable mutations.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients whose therapy is altered based upon the results of molecular testing.

II. To evaluate the percent of patients for which a local protocol offers a potential therapeutic option.

III. To evaluate the number of patients who are treated based on therapy guided by molecular profiling.

TERTIARY OBJECTIVES:

I. To compare the outcomes of patients treated with early therapy based on gene profiling with the outcomes of those treated via National Cancer National Comprehensive Cancer Network (NCCN) guideline recommended therapies (systemic therapy, liver directed therapy, hepatic resection) or expectant observation via measurement of progression free survival (PFS), via radiographic response rates, and via biochemical response rate.

II. To evaluate the prognostic power of commonly (>= 10%) detected mutations. III. To evaluate the impact of mammalian target of rapamycin (mTOR) pathway alterations (mutations of phosphatase and tensin homolog gene [PTEN], phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha [PIK3CA]) on efficacy of mTOR targeted therapeutics, as assessed by progression free survival (PFS) and response rate (RR).

IV. To evaluate the impact of o-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) status on the efficacy of an alkylating based chemotherapy regimen (Temodar, dacarbazine, streptozocin), as assessed by progression free survival (PFS) and response rate (RR).

V. To evaluate the impact of thymidine phosphorylase (TP) status on the efficacy of a fluoropyrimidine-based chemotherapy regimen (capecitabine, 5-fluorouracil), as assessed by progression free survival (PFS) and response rate (RR).

VI. To evaluate the impact of excision repair cross-complementing 1 (ERCC-1) status on the efficacy of a platinum-based chemotherapy regimen (carboplatin, cisplatin, oxaliplatin), as assessed by progression free survival (PFS) and response rate (RR).

OUTLINE:

Previously collected tissue samples are analyzed via mutational sequencing and immunohistochemistry.

After completion of study, patients are followed for up every 3-6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed neuroendocrine tumor which is metastatic, locally advanced or otherwise incurable (of any grade or primary site, excluding small cell lung cancers, large cell lung cancers, and Merkel cell carcinomas)
* Evaluable disease by radiographic imaging
* Adequate available tumor tissue (formalin-fixed paraffin-embedded [FFPE] tissue or cytologic material) for sequencing (containing > 50% tumor cellularity by histopathology) or consent to tumoral biopsy for fresh tissue; adequacy will be determined by our pathology department, under supervision of Dr. Gustafson
* Ability to understand and willingness to sign a written informed consent and Health Information Portability and Accountability Act (HIPAA) consent document
* Life expectancy of >= 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2

Exclusion Criteria:

* Localized neuroendocrine tumor for which the patient is eligible for a potentially curative surgical intervention
* Primary diagnosis of pulmonary small cell carcinoma, pulmonary large cell carcinoma or Merkel cell carcinoma
* Inability to provide informed consent
* Inadequate tissue available for genetic testing
* Any secondary active malignancy, excluding non-melanoma skin cancers; if the patient's prognosis will be primarily determined by their neuroendocrine tumor, the secondary malignancy is to be discounted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incurable neuroendocrine tumors, excluding small cell/large cell lung cancers and Merkel cell carcinomas
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-10-16 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2020-11-16 (Estimated)

PRIMARY OUTCOMES:
Feasibility, defined as the true proportion of patients whose CancerCode sequencing results in the identification of at least 1 actionable mutation | Up to 3 years

SECONDARY OUTCOMES:
Response rate, defined as at least a 30% decrease in target lesions when measureable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | Up to 3 years
  The response rate (with 95% two-sided confidence intervals) will be computed for all Arm B patients and separately for pre-specified subgroups (e.g., molecular profile-based treatment vs. NCCN guideline recommended).
Progression-free survival | Up to 3 years
  Progression-free survival time will be characterized for all Arm B patients and separately for pre-specified subgroups (e.g., molecular profile-based treatment vs. NCCN guideline recommended) using the method of Kaplan and Meier.
Overall survival | Up to 3 years
  Overall survival time will be characterized for all Arm B patients and separately for pre-specified subgroups (e.g., molecular profile-based treatment vs. NCCN guideline recommended) using the method of Kaplan and Meier.
Proportion of Arm B patients whose therapy is changed as a result of physician access to CancerCode results | Up to 3 years
Proportion of Arm B patients for whom a local protocol offers a potential therapeutic option based on CancerCode results | Up to 3 years

OTHER OUTCOMES:
Mutations occurring in greater than or equal to 10% of patients | Up to 3 years
  Log-rank test and Kaplan-Meier plots will be used to assess the relationships between progression free interval and common mutations (>= 10%) or immunohistochemistry (IHC) test results in the entire population.
Mutations in the mTOR pathway | Up to 3 years
  Log-rank test and Fisher's exact tests will be used to assess the relationships between mutations in the mTOR pathway and progression free interval or response among Arm B patients treated with mTOR inhibitors.
Prognostic value of MGMT status among patients on alkylating agents | Up to 3 years
Prognostic value of ERCC1 for patients on platinum-based regimens | Up to 3 years
Prognostic value of TP for patients on fluoropyrimidine-based regimens | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Engstrom, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States